CLINICAL TRIAL: NCT06571799
Title: A 4-month, Single Arm Study Evaluating the Efficacy and Safety of BENEV Exosome Regenerative Complex+® Post SylfirmX® RF Microneedling to Promote Hair Growth in Healthy Men and Women With Self-perceived Thinning Hair
Brief Title: Study Evaluating the Efficacy and Safety of BENEV Exosome Regenerative Complex+ for Self-perceived Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: Benev Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNV-EXO-HAIR-01
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-08

CONDITIONS: Thinning Hair
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Open label study evaluating the efficacy and safety
Masking Description: Open label study evaluating the efficacy and safety
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BENEV Exosome Regenerative Complex+ (Other): BENEV Exosome Regenerative Complex+® post SylFirmX® RF microneedling procedure applied to the scalp monthly for 4 sessions.
  Interventions: Other: BENEV Exosome Regenerative Complex+

INTERVENTIONS:
Other: BENEV Exosome Regenerative Complex+ — BENEV Exosome Regenerative Complex+® is an intensive dual-action complex formulated to absorb quickly into the skin and scalp delivering the concentrated power of stem cell derived lyophilized exosomes, potent growth factors, peptides, coenzymes, minerals, amino acids and vitamins.

SUMMARY:
The goal of this clinical trial is to further substantiate the effectiveness and safety of BENEV Exosome Regenerative Complex+ post SylFirmX® RF microneedling procedure for self-perceived thinning hair in healthy men and women ages 18-65 over the course of four months. Participants will be asked to have treatments monthly for 4 sessions, attend a follow up appointment 4 weeks after the 4th session, have photos taken of their hair and answer questionnaires related to their thinning hair.

DETAILED DESCRIPTION:
Exosomes represent promising new regenerative medicine treatments for facial rejuvenation and to enhance other cosmetic procedures. Exosomes can provide effective treatment for skin rejuvenation, scar reduction, hyperpigmentation, and hair growth. This new technology can be used alone but are often combined with other older existing aesthetic treatments. Specifically the use of exosomes in hair loss, has been anecdotally observed, but treatment protocols remain elusive and not universally accepted. Since hair loss has a multifactorial etiology, and traditional treatments have limitations, we explore the use of adipose tissue stem cell derived lyophilized exosomes for novel addition to the armamentarium of options to reverse hair thinning or shedding.

Exosome is defined as a 30~200 nm endoplasmic reticulum that is secreted for cell-to-cell communication and plays an important role in influencing the microenvironment around cells. ExoSCRT™ is an innovative technology to separate and refine 0.1% pure exosomes from stem cells and helps the virtualization of natural skin energy by affecting skin cells effectively. BENEV Exosome Regenerative Complex+® is an intensive dual-action complex formulated to absorb quickly into the skin and scalp delivering the concentrated power of stem cell derived lyophilized exosomes, potent growth factors, peptides, coenzymes, minerals, amino acids and vitamins.

The purpose of this clinical research study is to further evaluate the efficacy and safety of BENEV Exosome Regenerative Complex+® post SylFirmX® RF microneedling procedure of the scalp for self-perceived thinning hair in thirty (30) healthy male and female subjects, ages 18-65 years of age over the course of four (4) months.

ELIGIBILITY:
Inclusion Criteria

Subjects meeting all of the following criteria will be eligible for study entry:

1. Healthy males and females of all Fitzpatrick Skin Types between 18 and 65 years of age.
2. Subjects must be willing to provide verbal understanding and sign an Informed Consent Form, HIPAA Form and Photography Release Form approved by the Institutional Review Board.
3. Subjects must be in general good health, as determined by the Investigator.
4. Subjects with self-perceived hair thinning as determined on initial study assessment by the Investigator (excluding patients with medically diagnosed telogen effluvium).
5. Subjects willing to undergo a brief physical exam to include height, weight, blood pressure, pulse, physical scalp exam and basic systems evaluation (Skin, Respiratory, Cardiovascular, Gastrointestinal, Endocrine, Neurological and Musculoskeletal systems) by the Investigator.
6. Subjects willing to not substantially change their current diet, medications, or exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, or exercise routine, the subject will need to notify the clinic as soon as possible.
7. Females of child bearing potential (FOCBP) must be willing to have a urine pregnancy test and practice effective contraception for the duration of the study. (Effective contraception is defined as stabilized on oral contraceptive for at least 3 months as of the start of the study, intrauterine device, condom with spermicide, diaphragm with spermicide, implant, NuvaRing®, injection, transdermal patch or abstinence.) Females on birth control pills must have taken the same type of pill for at least 3 months prior to entering the study and must not change type during the study. Those who have used birth control pills in the past must have discontinued usage at least 3 months prior to the start of the study. The initiation of birth control should not have been associated with the initiation of hair loss/thinning.
8. FOCBP must have a negative urine pregnancy test at the Baseline Visit.
9. Subjects willing to give a blood sample collected for routine laboratory analysis (Complete Blood Count and Comprehensive Metabolic Panel).
10. Subjects willing to have 2-D digital photography of the entire head/hair region for overall evaluation of general hair growth and quality by the Investigator.
11. Subjects willing to have digital trichoscopy photography of the target site areas on the scalp for analysis of hair counts and other hair measurements.
12. Subjects willing to have RF microneedling procedure of the scalp region followed by application of IP.
13. Subjects must be willing and able to complete and understand the rating questionnaires.
14. Subjects must maintain a consistent length, cut, style and color throughout the four (4) month study period.
15. Subjects who have color treated hair must be willing to have the color treatment performed at the same time interval prior to visits.
16. Subjects willing to maintain their normal hair shampooing frequency, use a mild non-medicated shampoo and conditioner for the duration of the study and attend visits with clean and dry hair (shampoo must be done 24 hours or more prior to the visit).
17. Subjects must be willing and able to attend all study visits and comply with the post procedure and lifestyle instructions.

Exclusion Criteria

Subjects meeting any of the following criteria will be excluded from the study:

1. Subjects who are pregnant, nursing mothers, planning a pregnancy during the course of the study, or become pregnant during the study.
2. Subjects who have had a hair transplant.
3. Subjects with any known allergy or sensitivity to any shampoo and/or conditioner.
4. Subjects with known stressful incident within the last six months (e.g. death in family, miscarriage).
5. Subjects who have recently (within the last 3 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (3 months or longer) in order to be eligible for the study.
6. Subjects using Low Level Laser Therapy (LLLT) or other light therapy to treat thinning hair in the last 3 months.
7. Subjects who have regularly used Rogaine (Minoxidil), Nioxin and /or Finasteride or undergone any other hair or scalp treatments within the last 3 months.
8. Subjects who have used prescription drugs known to affect the hair growth cycle within the last 3 months (e.g., hormone-based birth control for less than 3 months, cyproterone acetate, aldactone/spironolactone or any 5-alpha-reductase inhibitor).
9. Subjects who have regularly used anti-androgenic therapies (i.e. spironolactone, flutamide, cyproterone acetate, progesterone and/or bicalutamide) or undergone any other hair or scalp treatments within the last 3 months.
10. Subjects suffering from other hair loss disorders, such as alopecia areata, scarring alopecia, androgenetic alopecia and telogen effluvium as determined during initial study assessment and physical exam by the Investigator.
11. Subjects with self-reported uncontrolled diseases (i.e. diabetes, hypertension, hyperthyroidism, hypothyroidism, etc.). Whether medical conditions are under control with or without treatment will be assessed on an individual basis by the Investigator based on her medical and clinical expertise.
12. Subjects with self-reported active hepatitis, immune deficiency, HIV or autoimmune disease.
13. Subjects having a known active dermatologic condition of the scalp that may place the subject at a greater risk or interfere with clinical evaluations (ie. seborrheic dermatitis, psoriasis, atopic dermatitis, advanced skin cancer, etc.) as determined by the Investigator based on her medical and clinical expertise.
14. Subjects who are unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function.
15. Subjects with any underlying disease that the Investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study.
16. Subjects with use of any medications that are known to potentially cause hair loss or affect hair growth as determined by the Investigator based on her medical and clinical expertise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Change in Terminal Hair Counts | Baseline to Day 120 or End of Study Visit
  Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of 40 micrometers. This is calculated by the Canfield HairMetrix System.
Change in Vellus Hair Counts | Baseline to Day 120 or End of Study Visit
  Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers. This is calculated by the Canfield HairMetrix System.
Change in Total Hair Counts | Baseline to Day 120 or End of Study Visit
  Total hairs equals the sum of Terminal and Vellus hairs in the target area. This is calculated by the Canfield HairMetrix System.

SECONDARY OUTCOMES:
Change in Terminal to Vellus Hair Count Ratio | Baseline to Day 120 or End of Study Visit
  Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of 40 micrometers. Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers. This ratio is calculated by the Canfield HairMetrix System.
Change in average hairs per follicular unit | Baseline to Day 120 or End of Study Visit
  This is the average number of hairs measured in each follicular unit.This is calculated by the Canfield HairMetrix System.
Change in average hair width | Baseline to Day 120 or End of Study Visit
  This is the average hair width calculated in micrometers by the Canfield HairMetrix System.
Change in follicular hair units per cm2 | Baseline to Day 120 or End of Study Visit
  This is the number of follicles per cm2 measured by the Canfield HairMetrix System.
Change in inter-follicular hair mean distance | Baseline to Day 120 or End of Study Visit
  This is the distance between hair follicles measured in millimeters by theCanfield HairMetrix System.
Change in Investigator Hair Growth Global Improvement Scale | Baseline to Day 120 or End of Study Visit
  The treating Investigator will complete this assessment by circling the number on the scale that corresponds to the description that best fits the current global growth improvement at delinated visits as indicated in the schedule of events, compared to baseline. The Investigator will complete this assessment during the study at Visits 2, 3, 4 and 5. The Investigator must complete this assessment using global photographs obtained compared to baseline. In addition, the Investigator may use their clinical judgment from the in-person visit.
  * 3 Greatly worsened
  * 2 Moderately worsened
  * 1 Slightly worsened 0 No change
    * 1 Slightly improved
    * 2 Moderately improved
    * 3 Greatly improved
Change in Investigator Hair Quality Global Improvement Scale | Baseline to Day 120 or End of Study Visit
  The treating Investigator will complete this assessment by circling the number on the scale that corresponds to the description that best fits the current hair quality at delinated visits as indicated in the schedule of events, as compared to the subject's hair quality at baseline. Assessment grading is to be based upon the Investigator's appraisal of hair brittleness, dryness, texture, shine, scalp coverage and overall appearance. The Investigator will complete this assessment during the study at Visits 2, 3, 4 and 5. The Investigator must complete this assessment using global photographs obtained compared to baseline. In addition, the Investigator may use their clinical judgment from the in-person visit.
  * 3 Greatly worsened
  * 2 Moderately worsened
  * 1 Slightly worsened 0 No change
    * 1 Slightly improved
    * 2 Moderately improved
    * 3 Greatly improved
Change in Hair Shedding Pull Test scores | Baseline to Day 120 or End of Study Visit
  The hair pull test will be performed by the Investigator to evaluate hair shedding. In the hair pull test, gentle traction will be applied on a group of hairs (approximately 60 hairs) from proximal to distal end, in the vertex area, both parietal areas and occipital area of the scalp. The grasp is made with the help of the thumb, index finger and middle finger, ensuring consistent pressure with each pull. If more than 10% (~6 or more) hairs come out with every pull, the test is considered positive. Subjects will be instructed not to shampoo or wash their hair 24 hours prior to the test for accurate results.
Change in Subject Hair Self-Assessment Questionnaire scores | Baseline to Day 120 or End of Study Visit
  This scale is used to rate the qualities listed below:
  1. Greatly Decreased/Worsened
  2. Moderately Decreased/Worsened
  3. Slightly Decreased/Worsened
  4. No Change
  5. Slightly Increased/Improved
  6. Moderately Increased/ Improved
  7. Greatly Increased/ Improved
  Overall hair growth Overall hair volume Scalp coverage Hair thickness Hair Fullness Hair quality Hair shine Hair strength Hair softness Amount of noticeable new hair Hair growth rate Hair growth on top of your head (scalp coverge) Hair growth of the hairline (at the front of your head or hairline coverage) Hair length (ability to grow longer than usual) Ease of styling Overall hair appearance Nail Strength Nail Growth Rate Growth of Eyebrow Hair Growth of Eyelashes Skin Smoothness Overall Skin Health
Change in Hair Treatment Subject Satisfaction Questionnaire scores | Baseline to Day 120 or End of Study Visit
  1. How satisfied are you with this treatment for your thinning hair? 5 = Very Satisfied 4 = Satisfied 3 = Neutral 2 = Dissatisfied 1 = Very Dissatisfied
  2. How satisfied are you with the overall health of your hair after this treatment? 5 = Very Satisfied 4 = Satisfied 3 = Neutral 2 = Dissatisfied 1 = Very Dissatisfied
  3. Overall, how satisfied are you with the ease of this treatment? 5 = Very Satisfied 4 = Satisfied 3 = Neutral 2 = Dissatisfied 1 = Very Dissatisfied
  4. Overall, now that you have tried this treatment and completed the study, how likely are you to continue the treatment in the future? 5 = Very Likely 4 = Somewhat Likely 3 = Neutral 2 = Somewhat Unlikely 1 = Very Unlikely
  5. Overall, how likely are you to recommend this treatment to a family member or friend? 5 = Very Likely 4 = Somewhat Likely 3 = Neutral 2 = Somewhat Unlikely 1 = Very Unlikely

OTHER OUTCOMES:
Frequency of both local and systemic Adverse Events | Baseline to Day 120 or End of Study Visit
  An adverse event is any adverse change from the subject's baseline condition, i.e. any subjective signs and symptoms, or change in a concomitant disease present at the screening visit. This includes inter-current signs, symptoms, illness and significant deviations from baseline which may occur during the course of the clinical study, whether considered related to treatment or not.
Changes in Clinical laboratory analyses of Complete Blood Count without Differential and with Platelets | Baseline to Day 120 or End of Study Visit
  Number of participants with abnormal clinical laboratory analyses of Complete Blood Count with Differential and with Platelets Panel (this is a single blood panel). The analyses will be conducted on blood samples collected from subjects at Baseline and Day 120 visits. All results will be reported, including results that are abnormal. The Complete Blood Count with Differential and with Platelets Panel (single blood panel) contains the following tests: WBC, RBC,Hemoglobin, Hematocrit, MCV, MCH, MCHC, RDW, Platelets
Change in Clinical laboratory analyses of Complete Metabolic Panel | Baseline to Day 120 or End of Study Visit
  Number of participants with abnormal clinical laboratory analyses of Complete Metabolic Panel (this is a single blood panel). The analyses will be conducted on blood samples collected from subjects at Baseline and Day 120 visits. All results will be reported, including results that are abnormal. The Complete Metabolic Panel includes the following tests:alkaline phosphatase(ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, blood urea nitrogen (BUN), creatinine, sodium, potassium, carbon dioxide, chloride, albumin, total protein, glucose, and calcium

CONTACTS AND LOCATIONS:
Locations (1):
- Ablon Skin Institute & Research Center, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ablon G. An Exosome Regenerative Complex Plus Microneedling Promotes Hair Growth in Subjects With Self-Perceived Thinning Hair. J Drugs Dermatol. 2025 Oct 1;24(10):988-994. doi: 10.36849/JDD.9244. PMID 41037530